CLINICAL TRIAL: NCT04690985
Title: Dietary Behaviour Change Intervention on Managing Sarcopenic Obesity in Community-dwelling Older People: a Feasibility and Pilot Study
Brief Title: Dietary Behaviour Change Intervention Among Older People With Sarcopenic Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr. Justina Liu Yat Wa, Associate Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20191007001
Record Dates: First submitted 2020-10-19; First posted 2020-12-31 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Sarcopenic Obesity
Keywords: dietary behaviour change; sarcopenic obesity; community; randomized controlled trial

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Sham Comparator): The control group will be asked to continue their own daily routes. One research assistant, who will not be involved in other procedures of the study, will contact with the participants to talk about different issues except the SO related topic. The frequency of face-to-face meetings and telephone calls will be similar to the experimental group. The issues talked in the control group could be as follows but not limited: a) normal social communication topics such as greetings, recent living conditions, news in the past week; b) health consultations asked by the participants; c) avoid to mention dietary or exercise related information. An appointment of post-test will be made in the last time telephone call.
  Interventions: Other: Social contact
- Experimental group (Experimental): The experimental group will be required to adhere to a diet consisting of a 12% reduction in calorie and a 1.2-1.5 g/kg body weight/day intake of protein. The participants will receive 6 times face-to-face meetings (on week 1, 2, 3, 4, 8 and 12) and weekly telephone call. Each face-to-face meetings will last for around 1 hour, during which the reseacher will help to establish the participants' intention for dietary behavior change, then help transform the intention into detailed plan, and help monitor the execution of the plan continuously.
  Interventions: Behavioral: Dietary behaviour change

INTERVENTIONS:
Behavioral: Dietary behaviour change — The intervention consists of dietary guidance and behaviour change techniques, which will last for 15 weeks. The experimental group will be required to adhere to a diet consisting of a 12% reduction in calorie and a 1.2-1.5 g/kg body weight/day intake of protein. The participants will receive the dietary behaviour change guidance in 6 times face-to-face meetings and weekly telephone calls. They will also be asked to take daily food diary.
  Arms: Experimental group
Other: Social contact — The control group will not be required any dietary changes. The investigator will contact with the control group with the same frequency and numbers of experimental group. But the chat topic will not be related to sarcopenic obesity or dietary guidance.
  Arms: Control group

SUMMARY:
The aim of this study is to evaluate the feasibility and preliminary effects of dietary behavior change intervention on the management of sarcopenic obesity (SO) among older people in the community.

The feasibility and preliminary effects of the intervention will be tested using a two-armed pilot randomized controlled trial among older people (N=60) with SO in the community in Nanjing, China. Finally, 10 participants will be invited to join a semi-structured interview to explore their perceptions about the whole intervention process.

It is hypothesized that the experimental group will have a greater improvement in the body composition, muscle strength and physical function compared to the control group after receiving the 15-week dietary behavior change intervention.

DETAILED DESCRIPTION:
The pilot study is a single-blind, two-arm randomized controlled trial. A total of 60 subjects (60 years old or more) are planned to be recruited. The subjects will be randomly divided into 2 groups witht a ratio of 1:1. One is the experimental group and the other is the control group.

The experimental group will receive 15 weeks of dietary intervention, including 6 face-to-face meetings and weekly telephone call. Each meeting lasts for 1 hour. The participants in the experimental group are required to control of calorie intake (decrease energy intake by 12%) and increase protein intake (1.2-1.5 g/body weight kg/day), and take dietary diary.

The control group will not receive any dietary interventions. They will only receive regular contacts with a similar frequency as the experimental group. The content of the conversations will not involve any topics related to SO.

After the intervention, 10-15 people from the experimental group will be randomly selected to receive semi-structured individual interview, which will last around 1 hour. The researcher plan to understand their feelings about participating in the study.

ELIGIBILITY:
Inclusion Criteria:

* community-dwelling older people aged 60 years old or above;
* handgrip strength < 28 kg for men and < 18 kg for women;
* BMI ≥ 28% or waist circumference ≥ 85 cm in men and ≥ 80 cm in women;
* be able to read and write without severe hearing and vision problems.

Exclusion Criteria:

* suffering from severe heart disease or metabolic disorders (e.g. renal diseases, diabetes) or autoimmune disease, cancer, or any other diseases/ conditions which may affect food intake and digestion or amputee;
* cognitively impaired (e.g. dementia) may impede the delivery of the intervention;
* under special diet restriction such as on diabetes disease diet, vegetarian, ketogenic diet, etc.;
* using of medications that may influence eating behavior, digestion or metabolism (such as weight loss medication);
* addicted to alcohol;
* a metal device is implanted in the body;
* be engaged in another trials.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Changes of muscle strength | Change from baseline to 1 week after the programme
  Handgrip strength (kg) will be measured by using the jamar dynamometer.
Changes of physical function | Change from baseline to 1 week after the programme
  The Short Physical Performance Battery (SPPB) scale will be used to measure physical function, which is a well-established tool for monitoring function in older people, which contains three kinds of assessments: stand for 10 seconds with feet in 3 different positions, 3-meter or 4-meter walking speed test, and time to rise from a chair for five times. The scores of SPPB range from 0 (worst performance) to 12 (best performance).
Changes of skeletal muscle mass | Change from baseline to 1 week after the programme
  Skeletal muscle mass (kg) will be measured by using bioelectrical impedance analysis.
Changes of body weight | Change from baseline to 1 week after the programme
  Body weight (kg) will be measured.
Changes of fat mass | Change from baseline to 1 week after the programme
  Fat mass (kg) will be measured by using bioelectrical impedance analysis.
Changes of visceral fat score | Change from baseline to 1 week after the programme
  Visceral fat score will be measured by using bioelectrical impedance analysis. Maintain a visceral fat score below 10 means good health.
Changes of body mass index | Change from baseline to 1 week after the programme
  The weight and height will be combined to report BMI in kg/m^2.
Changes of percentage of body fat | Change from baseline to 1 week after the programme
  Percentage of body fat will be reported by the percent of body fat mass in whole body weight.
Changes of waist-to-hip ratio | Change from baseline to 1 week after the programme
  Waist circumference(cm) and hip circumference (cm) will be measured to report the waist-to-hip ratio.
Recruitment rate | Baseline
  The proportion of participants who consent to join the study over the eligible participants.
Attrition rate | At the end of the 15-week programme
  The percentage of participants who withdraw from the study and their reasons for withdrawing.
Adherence to diet regimen | Throughout the 15-week programme
  Diet adherence will be assessed by the session attendance (Rate of attendance in 6 sessions).
Occurrence of adverse events | Throughout the 15-week programme
  Any adverse events at home will be recorded.

SECONDARY OUTCOMES:
Mini Nutritional Assessment (MNA) Short-form | Change from baseline to 1 week after the programme
  Participants' nutritional status will be assessed through the Mini Nutritional Assessment (MNA). It is a simple and quick tool for assessing older people who are malnourished or at risk of malnutrition. The MNA Short-form contains 6 items. Questions are weighted, 2-3 ponits per item. Scores are categoried as 0-7 (malnourished), 8-11 (at risk of malnutrition), 12-14 (normal nutritional status).
Nutrition Self-efficacy Scale | Change from baseline to 1 week after the programme
  The nutrition self-efficacy scale is one part of the Health-Specific Self-efficacy Scale which was developed by Ralf Schwarzer and Britta Renner. The nutritional self-efficacy scale is a 5-item scale, and each item is rated on 4-point likert scale from 1= very uncertain, 2=rather uncertain, 3=rather certain, 4=very certain. Higher score means higher self-efficacy.
Dietary quality index-International | Change from baseline to 1 week after the programme
  The DQI-I will be used to estimate the dietary quality of participants. It is a well-used questionnaire without being affected by culture.
Short Form Health Survey (SF-36) | Change from baseline to 1 week after the programme
  The Short Form (36) Health Survey is a 36-item, patient-reported survey of patient health, which is always used to assess people's health status and quality of life. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability.
International Physical Activity Questionnaire Short-form (IPAQ-SF) | Change from baseline to 1 week after the programme
  The International Physical Activity Questionnaires Short-form (IPAQ-SF) contains (4 generic items, which is used to evaluate the vigorous activities that participants did in the last 7 days. MET minutes represent the amount of energy expended carrying out physical activity. The higher score means engaging in higher level of physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Justina Liu, PhD, Study Chair — The Hong Kong Polytechnic University; Yueheng Yin, PhD, Principal Investigator — The Hong Kong Polytechnic University; Maritta Valimaki, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- Jiangning Dongshan Community Healthcare Center, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
For confidentiality, the data will be kept anonymous and the information of all participants will be replaced by reference codes. The data collected will be kept in a locked place and electronic versions will be encrypted, and only be accessible by the researchers. All data will be destroyed within 3 years after the completion of this research.

REFERENCES:
- [Background] Anthony TG. Mechanisms of protein balance in skeletal muscle. Domest Anim Endocrinol. 2016 Jul;56 Suppl(Suppl):S23-32. doi: 10.1016/j.domaniend.2016.02.012. PMID 27345321
- [Background] Bergamini E, Cavallini G, Donati A, Gori Z. The anti-ageing effects of caloric restriction may involve stimulation of macroautophagy and lysosomal degradation, and can be intensified pharmacologically. Biomed Pharmacother. 2003 Jul-Aug;57(5-6):203-8. doi: 10.1016/s0753-3322(03)00048-9. PMID 12888255
- [Background] Beasley JM, Shikany JM, Thomson CA. The role of dietary protein intake in the prevention of sarcopenia of aging. Nutr Clin Pract. 2013 Dec;28(6):684-90. doi: 10.1177/0884533613507607. Epub 2013 Oct 25. PMID 24163319
- [Background] Bellg AJ, Borrelli B, Resnick B, Hecht J, Minicucci DS, Ory M, Ogedegbe G, Orwig D, Ernst D, Czajkowski S; Treatment Fidelity Workgroup of the NIH Behavior Change Consortium. Enhancing treatment fidelity in health behavior change studies: best practices and recommendations from the NIH Behavior Change Consortium. Health Psychol. 2004 Sep;23(5):443-51. doi: 10.1037/0278-6133.23.5.443. PMID 15367063
- [Background] Chen C, Lu FC; Department of Disease Control Ministry of Health, PR China. The guidelines for prevention and control of overweight and obesity in Chinese adults. Biomed Environ Sci. 2004;17 Suppl:1-36. No abstract available. PMID 15807475
- [Background] Chen LK, Woo J, Assantachai P, Auyeung TW, Chou MY, Iijima K, Jang HC, Kang L, Kim M, Kim S, Kojima T, Kuzuya M, Lee JSW, Lee SY, Lee WJ, Lee Y, Liang CK, Lim JY, Lim WS, Peng LN, Sugimoto K, Tanaka T, Won CW, Yamada M, Zhang T, Akishita M, Arai H. Asian Working Group for Sarcopenia: 2019 Consensus Update on Sarcopenia Diagnosis and Treatment. J Am Med Dir Assoc. 2020 Mar;21(3):300-307.e2. doi: 10.1016/j.jamda.2019.12.012. Epub 2020 Feb 4. PMID 32033882
- [Background] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jul 1;48(4):601. doi: 10.1093/ageing/afz046. No abstract available. PMID 31081853
- [Background] Goisser S, Kemmler W, Porzel S, Volkert D, Sieber CC, Bollheimer LC, Freiberger E. Sarcopenic obesity and complex interventions with nutrition and exercise in community-dwelling older persons--a narrative review. Clin Interv Aging. 2015 Aug 6;10:1267-82. doi: 10.2147/CIA.S82454. eCollection 2015. PMID 26346071
- [Background] Hertzog MA. Considerations in determining sample size for pilot studies. Res Nurs Health. 2008 Apr;31(2):180-91. doi: 10.1002/nur.20247. PMID 18183564
- [Background] Schwarzer R, Renner B. Social-cognitive predictors of health behavior: action self-efficacy and coping self-efficacy. Health Psychol. 2000 Sep;19(5):487-95. PMID 11007157
- [Background] Schwarzer R, Lippke S, Luszczynska A. Mechanisms of health behavior change in persons with chronic illness or disability: the Health Action Process Approach (HAPA). Rehabil Psychol. 2011 Aug;56(3):161-70. doi: 10.1037/a0024509. PMID 21767036
- [Background] Yin YH, Liu JYW, Valimaki M. Effectiveness of non-pharmacological interventions on the management of sarcopenic obesity: A systematic review and meta-analysis. Exp Gerontol. 2020 Jul 1;135:110937. doi: 10.1016/j.exger.2020.110937. Epub 2020 Mar 30. PMID 32240820
- [Background] Li L, Wang HM, Shen Y. Chinese SF-36 Health Survey: translation, cultural adaptation, validation, and normalisation. J Epidemiol Community Health. 2003 Apr;57(4):259-63. doi: 10.1136/jech.57.4.259. PMID 12646540
- [Background] Zhang CX, Ho SC. Validity and reproducibility of a food frequency Questionnaire among Chinese women in Guangdong province. Asia Pac J Clin Nutr. 2009;18(2):240-50. PMID 19713184
- [Background] Lee PH, Yu YY, McDowell I, Leung GM, Lam TH, Stewart SM. Performance of the international physical activity questionnaire (short form) in subgroups of the Hong Kong chinese population. Int J Behav Nutr Phys Act. 2011 Aug 1;8:81. doi: 10.1186/1479-5868-8-81. PMID 21801461
- [Background] Deutz NE, Bauer JM, Barazzoni R, Biolo G, Boirie Y, Bosy-Westphal A, Cederholm T, Cruz-Jentoft A, Krznaric Z, Nair KS, Singer P, Teta D, Tipton K, Calder PC. Protein intake and exercise for optimal muscle function with aging: recommendations from the ESPEN Expert Group. Clin Nutr. 2014 Dec;33(6):929-36. doi: 10.1016/j.clnu.2014.04.007. Epub 2014 Apr 24. PMID 24814383
- [Background] Fontana L, Klein S. Aging, adiposity, and calorie restriction. JAMA. 2007 Mar 7;297(9):986-94. doi: 10.1001/jama.297.9.986. PMID 17341713
- [Background] Kraus WE, Bhapkar M, Huffman KM, Pieper CF, Krupa Das S, Redman LM, Villareal DT, Rochon J, Roberts SB, Ravussin E, Holloszy JO, Fontana L; CALERIE Investigators. 2 years of calorie restriction and cardiometabolic risk (CALERIE): exploratory outcomes of a multicentre, phase 2, randomised controlled trial. Lancet Diabetes Endocrinol. 2019 Sep;7(9):673-683. doi: 10.1016/S2213-8587(19)30151-2. Epub 2019 Jul 11. PMID 31303390
- [Background] Morley JE, Argiles JM, Evans WJ, Bhasin S, Cella D, Deutz NE, Doehner W, Fearon KC, Ferrucci L, Hellerstein MK, Kalantar-Zadeh K, Lochs H, MacDonald N, Mulligan K, Muscaritoli M, Ponikowski P, Posthauer ME, Rossi Fanelli F, Schambelan M, Schols AM, Schuster MW, Anker SD; Society for Sarcopenia, Cachexia, and Wasting Disease. Nutritional recommendations for the management of sarcopenia. J Am Med Dir Assoc. 2010 Jul;11(6):391-6. doi: 10.1016/j.jamda.2010.04.014. PMID 20627179
- [Background] Newman AB, Lee JS, Visser M, Goodpaster BH, Kritchevsky SB, Tylavsky FA, Nevitt M, Harris TB. Weight change and the conservation of lean mass in old age: the Health, Aging and Body Composition Study. Am J Clin Nutr. 2005 Oct;82(4):872-8; quiz 915-6. doi: 10.1093/ajcn/82.4.872. PMID 16210719
- [Background] Zhang CQ, Zhang R, Schwarzer R, Hagger MS. A meta-analysis of the health action process approach. Health Psychol. 2019 Jul;38(7):623-637. doi: 10.1037/hea0000728. Epub 2019 Apr 11. PMID 30973747
- [Derived] Yin YH, Liu JYW, Valimaki M. Dietary behaviour change intervention for managing sarcopenic obesity among community-dwelling older people: a pilot randomised controlled trial. BMC Geriatr. 2023 Sep 26;23(1):597. doi: 10.1186/s12877-023-04327-w. PMID 37752447

DOCUMENTS (1):
  • Informed Consent Form (2019-10-15): https://cdn.clinicaltrials.gov/large-docs/85/NCT04690985/ICF_000.pdf